CLINICAL TRIAL: NCT02025725
Title: Phase 3 Study of Intranasal Metoclopramide in Women With Symptomatic Diabetic Gastroparesis
Brief Title: Multicenter Study to Evaluate the Efficacy and Safety of Metoclopramide Nasal Spray in Women With Diabetic Gastroparesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evoke Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: METO-IN-003
Record Dates: First submitted 2013-12-29; First posted 2014-01-01 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Gastroparesis
Keywords: Gastroparesis; Diabetic; Delayed gastric emptying; Gastric stasis; Nausea; Vomiting; Bloating; Abdominal pain; Early satiety; Gastropathy
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Abdominal Pain; Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 mg Metoclopramide Nasal Spray (Experimental): Metoclopramide Nasal Spray 10 mg, 30 minutes before meals and at bedtime (QID) for 4 weeks
  Interventions: Drug: Metoclopramide Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): Placebo Nasal Spray 30 minutes before meals and at bedtime (QID) for 4 weeks
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Metoclopramide Nasal Spray — nasal spray formulation of metoclopramide
  Other Names: EVK-001
  Arms: 10 mg Metoclopramide Nasal Spray
Drug: Placebo Nasal Spray — nasal spray formulation with vehicle only
  Other Names: EVK-001 Placebo
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is provide confirmation of the safety and efficacy of Metoclopramide Nasal Spray compared to placebo in reducing the symptoms of diabetic gastroparesis in adult women.

DETAILED DESCRIPTION:
Diabetic women with clinical symptoms attributed to diabetic gastroparesis and documentation of delayed gastric emptying who meet the protocol-specified entry criteria will be randomized to Metoclopramide Nasal Spray 10 mg or placebo administered as a single intranasal spray four (4) times daily; 30 minutes before meals and at bedtime for a total of four (4) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant, non lactating female subjects between the ages of 18 and 75 years
* Willingness and ability to give written informed consent
* The ability to read, understand and speak English
* Prior diagnosis of Type 1 or Type 2 diabetes
* Diagnosis of diabetic gastroparesis with confirmation of delayed gastric emptying
* A mean daily gastroparesis symptom score of ≥1.4 and ≤3.5 prior to randomization
* Subjects of childbearing potential must agree to use contraception
* Willingness to discontinue current treatment for diabetic gastroparesis and to avoid all proscribed (excluded) medications, as specified by the protocol, for the duration of the study

Exclusion Criteria:

* Gastric bypass, gastric banding, gastric pacemaker, post surgical causes of gastroparesis and disorders known to be associated with abnormal gastrointestinal motility
* A history of allergic or adverse responses, including, but not limited to, acute dystonic reactions and tardive dyskinesia, to metoclopramide or any comparable or similar product
* A history of, or physical findings suggestive of, tardive dyskinesia
* A history of epilepsy or currently using and unwilling or unable stop other drugs known to be associated with extrapyramidal reactions at screening
* A history of allergy to any of the ingredients in the study drug formulation
* A history of organ transplant, chronic pancreatitis, gross malabsorptive syndromes, celiac disease, active inflammatory bowel disease (IBD), or symptomatic irritable bowel syndrome (IBS)
* Malignancy (with the exception of treated squamous cell or basal cell carcinoma of the skin) currently present, initially diagnosed or recurring within five (5) years of screening
* Renal dysfunction calculated as creatinine clearance (CrCl) <40 mL/min at screening
* Hemoglobin A1c >11.5% at screening
* Subjects who are trying to conceive, are pregnant, or are lactating

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-03-27; Primary Completion 2016-05-27 (Actual); Study Completion 2016-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn R. Carlson, DMD, MD, Study Director — Evoke Pharma, Inc.
Locations (50):
- United States (50):
  - Birmingham Gasteroenterology Associates, P.C., Birmingham, Alabama
  - Digestive Specialists of the Southeast, Dothan, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Central Arizone Medical Associates/Clinical Research Advantage, Mesa, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Precision Research Institute, LLC, Chula Vista, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Precision Research Institute, LLC, San Diego, California
  - The Center for Gastrointestinal Disorders, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - International Research Associates, LLC, Miami, Florida
  - Advanced Medical Research, Port Orange, Florida
  - Tri-County Research, Athens, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Newton Medical Center, Conyers, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Indiana University Health UH 1634, Indianapolis, Indiana
  - Professional Research Network of Kansas, Wichita, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Gastrointestional Associates, Jackson, Mississippi
  - Kansas City Gastroenterology & Hepatology, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Premier Medical Group of the Hudson, PC, Poughkeepsie, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - LeBauer Research Associates, Greensboro, North Carolina
  - Kinston Medical Specialist Clinical Research Office, Kinston, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Dayton Gastroenterology, Beavercreek, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Lovelace Scientific Resources, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Burke Internal Medicine, Burke, Virginia
  - Manassas Clinical Research, Manassas, Virginia
  - National Clinical Research, Norfolk, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCallum RW, Parkman HP, Fass R, Bhandari BR, Carlson MR, Buck RD. Metoclopramide Nasal Spray in Women With Symptomatic Diabetic Gastroparesis: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study. Clin Gastroenterol Hepatol. 2024 Dec;22(12):2497-2505.e5. doi: 10.1016/j.cgh.2023.10.022. Epub 2023 Nov 2. PMID 37924856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 27 March 2014 to 27 May 2016
  Types of Location: Medical Clinics, University-Based Practices
  Screening Period consisted of Washout Period, Qualification Period and Baseline Period. Mean daily Gastroparesis Symptom Assessment (GSA) total score ≥ 1.4 and ≤ 3.5 was required during Qualification and Baseline periods
Pre-assignment Details: 613 participants Screened, 205 participants completed and randomized to treatment.
  Negative Gastric Emptying Scintigraphy 129 Inclusion/Exclusion Failed 213 Withdrawal by participant 25 Other Reasons 41
Period: Overall Study
Arm/Group | 10 mg Metoclopramide Nasal Spray | Placebo Nasal Spray
Started | 102 | 103
Completed | 91 | 99
Not Completed | 11 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Post-dose QTcB > 270 msec | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Metoclopramide Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Categorical [Count of Participants; unit: Participants]
  Age (years): <=18 years | 0 | 0 | 0
  Age (years): Between 18 and 65 years | 87 | 90 | 177
  Age (years): >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (11.6) | 52.5 (10.9) | 52.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Only females were enrolled in this study
  Participants
    Female | 102 | 103 | 205
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 91 | 89 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race categories may add to > 100% since a subject's eCRF could indicate multiple races.
  Participants
    American Indian or Alaska Native | 2 | 3 | 5
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 20 | 37 | 57
    White | 78 | 63 | 141
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 103 | 205
Qualification Mean Daily GSA Score [Mean (Standard Deviation); unit: units on a scale] | 2.259 (0.481) | 2.242 (0.487) | 2.251 (0.483)
Baseline Mean Daily GSA Score [Mean (Standard Deviation); unit: units on a scale] | 2.28 (0.518) | 2.30 (0.552) | 2.29 (0.53)
Diabetes Mellitus Type [Count of Participants; unit: Participants]
  Type 1 | 13 | 11 | 24
  Type 2 | 89 | 92 | 181
Diabetes Mellitus Duration [Mean (Standard Deviation); unit: years] | 12.4 (10.51) | 13.4 (10.9) | 12.9 (10.7)
Current Diabetes Mellitus Treatment [Count of Participants; unit: Participants]
  Diet | 30 | 33 | 63
  Oral Diabetic Medications | 69 | 74 | 143
  Insulin | 51 | 54 | 105
  Other | 11 | 17 | 28
  None | 0 | 1 | 1
Co-Existing Complications of Diabetes [Count of Participants; unit: Participants]
  No Complications | 64 | 60 | 124
  Any Complication | 38 | 41 | 79
  Diabetic Retinopathy | 7 | 2 | 9
  Neuropathy | 35 | 39 | 74
  Nephropathy | 2 | 1 | 3
  Peripheral Vascular Disease/Amputation | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Gastroparesis Symptom Assessment (GSA), a Patient Reported Outcome Measure
Description: Change from the Baseline Period to Week 4 of the Treatment Period in the mean daily Gastroparesis Symptom Assessment (GSA) total score for subjects receiving Metoclopramide Nasal Spray 10 mg versus subjects receiving placebo. The GSA minimum value is 0 (no symptoms) and the maximum value is 4 (very severe symptoms). A higher score is a worse outcome.
Time Frame: Baseline Period to Week 4 of the Treatment Period
Population: Intent-to-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 10 mg Metoclopramide Nasal Spray: Metoclopramide Nasal Spray 10 mg, 30 minutes before meals and at bedtime for 4 weeks
  Metoclopramide Nasal Spray: nasal spray formulation of metoclopramide
- Placebo Nasal Spray: Placebo Nasal Spray 30 minutes before meals and at bedtime for 4 weeks
  Placebo Nasal Spray: nasal spray formulation with vehicle only
Arm/Group | 10 mg Metoclopramide Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 102 | 103
score on a scale | -0.925 (0.935) | -0.896 (0.947)
Statistical Analysis 1: Comparison: 10 mg Metoclopramide Nasal Spray vs Placebo Nasal Spray; Test type: Superiority; p = 0.881, ANCOVA

2. Post Hoc Outcome: Gastroparesis Symptom Assessment (GSA)
Description: Change from the Baseline Period to Weeks 1, 2, 3 and 4 of the Treatment Period in the mean daily Gastroparesis Symptom Assessment (GSA) total score in subjects with moderate to severe symptoms at Baseline (GSA score greater than 2.7) receiving Metoclopramide Nasal Spray 10 mg versus subjects receiving placebo. The GSA minimum value is 0 (no symptoms) and the maximum value is 4 (very severe symptoms). A higher score is a worse outcome.
Time Frame: Baseline Period to Weeks 1, 2, 3 and 4 of the Treatment Period
Population: Subjects in the intent-to-treat population with moderate to severe disease (symptoms) at Baseline (i.e., baseline GSA scores higher than 2.7 on the 0-4 scale). Results presented are Weeks 1, 2, 3 and 4 compared to the Baseline Period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 10 mg Metoclopramide Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 52 | 53
score on a scale
  Week 1 of Treatment compared to Baseline Period | -0.587 (0.520) | -0.388 (0.444)
  Week 2 of Treatment compared to Baseline Period | -0.949 (0.864) | -0.616 (0.635)
  Week 3 of Treatment compared to Baseline Period | -1.095 (0.912) | -0.750 (0.785)
  Week 4 of Treatment compared to Baseline Period | -1.218 (0.991) | -0.857 (0.938)
Statistical Analysis 1: Comparison: 10 mg Metoclopramide Nasal Spray vs Placebo Nasal Spray; Change in mean daily GSA total score from Baseline to Week 1: metoclopramide nasal spray minus placebo; Test type: Superiority; p = 0.036, ANCOVA; Mean Difference (Net) = -0.201
Statistical Analysis 2: Comparison: 10 mg Metoclopramide Nasal Spray vs Placebo Nasal Spray; Change in mean daily GSA total score from Baseline to Week 2: metoclopramide nasal spray minus placebo; Test type: Superiority; p = 0.025, ANCOVA; Mean Difference (Net) = -0.336
Statistical Analysis 3: Comparison: 10 mg Metoclopramide Nasal Spray vs Placebo Nasal Spray; Change in mean daily GSA total score from Baseline to Week 3: metoclopramide nasal spray minus placebo; Test type: Superiority; p = 0.039, ANCOVA; Mean Difference (Net) = -0.347
Statistical Analysis 4: Comparison: 10 mg Metoclopramide Nasal Spray vs Placebo Nasal Spray; Change in mean daily GSA total score from Baseline to Week 4: metoclopramide nasal spray minus placebo; Test type: Superiority; p = 0.085, ANCOVA; Mean Difference (Net) = -0.364

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected through the last study visit (Day 28). Serious AEs (SAEs) were collected for up to 30 days after the final dose of study drug.
Description: Adverse event (AE) collection began after subjects signed the Informed Consent Form and continued until the subject was discharged from the study due to completion or Early Termination. All AEs observed by the Investigator, reported by the subject, from laboratory findings, or other means, were collected. AEs after the first dose of study drug were classified as treatment-emergent AEs.
Arm/Group | 10 mg Metoclopramide Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/103
Serious Adverse Events (participants affected / at risk) | 3/102 | 2/103
Other Adverse Events (participants affected / at risk) | 21/102 | 36/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg Metoclopramide Nasal Spray (N=102) | Placebo Nasal Spray (N=103)
orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
chalazion (Eye disorders) | 1 (1) | 0 (0)
anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg Metoclopramide Nasal Spray (N=102) | Placebo Nasal Spray (N=103)
Headache (Nervous system disorders) | 5 (6) | 7 (9)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less